CLINICAL TRIAL: NCT05453734
Title: The Effect of Progressive Muscle Relaxation Exercises on Breastfeeding Self-Efficacy and Depression Level of Mothers With Preterm Infants: A Randomized Controlled Study
Brief Title: The Effect of Progressive Muscle Relaxation Exercises
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Kadriye Sahin, Research Assistant in the Department of Child Health and Diseases Nursing, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: SHN503434
Record Dates: First submitted 2022-06-22; First posted 2022-07-12 (Actual); Last update posted 2022-07-12 (Actual); Status verified 2022-07

CONDITIONS: Preterm; Mothers
Keywords: mother; self efficacy; postpartum depression; preterm infant; progressive muscle relaxation
MeSH Terms: conditions — Premature Birth; Depression, Postpartum

STUDY DESIGN:
Intervention Model Description: Randomized controlled experimental design
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group: The group applied Progressive Muscle Relaxation Exercises (Experimental): Introductory information form and EPDS were completed by the mothers before the PMR exercises. PMR exercises were applied and training was given to the mothers by the researcher in the milking room (a quiet room) located on the NICU floor (approximately 40 minutes). The application was continued until the mother was able to do the PMR exercises on her own. After the application and training, the mother was given guidance on PMR. The mother was asked to perform the exercises twice a day, in the morning and evening, and record them on the follow-up form. The researcher's contact number was given to the mother for counseling in case she had difficulty following the steps of the PMR exercises. During the follow-ups, the mother was called by the researcher and a message was sent to ensure her continuity in the exercises. At the end of the 1st and 2nd weeks of the follow-up, BSES, EPDS and patient follow-up forms were filled when the mother came for routine controls.
  Interventions: Procedure: Progressive Muscle Relaxation Exercises
- Control group: The group without any ıntervention (No Intervention): Introductory information form, the BSES, and the EPDS were initially applied to the mothers. At the end of the 1st and 2nd weeks of the follow-up, the BSES and the EPDS were applied to the mothers. At the end of the 2nd week, it was told the mothers how to practice the PMR exercises and the guideline on the PMR exercises was given to them.

INTERVENTIONS:
Procedure: Progressive Muscle Relaxation Exercises — Before data collection, one of the researchers received training and certification from a psychotherapist specialist in this field to be able to apply the PMR exercises. The guidelines on the PMR exercises were prepared in line with the literature and training received by the researcher. In the guidelines, the person is asked to be in a comfortable place and position, to reach the face by following the large muscle groups gradually, starting from the feet, to tense the muscles in each step, and then to release them. It is necessary to take a deep breath after each muscle group, to stop for a while, and release it slowly
  Arms: Experimental Group: The group applied Progressive Muscle Relaxation Exercises

SUMMARY:
Purpose This study was carried out to examine the effectiveness of Progressive Muscle Relaxation (PMR) exercises on mothers' breastfeeding self-efficacy and depression level with preterm infants.

Methods This study was conducted in a randomized controlled experimental design. The sample of the study consisted of 70 mothers with 32-36 weeks preterm infants (35/35 in experimental/control group) and hospitalized in the Neonatal Intensive Care Unit (NICU) of the university hospital in which the study was conducted. Introductory information form; Breastfeeding Self-Efficacy Scale (BSES), Edinburgh Postpartum Depression Scale (EPDS), and patient follow-up form were used to collect data. Progressive Muscle Relaxation (PMR) exercises were practiced on the mothers in the experimental group. The mothers were given training and instructions about the exercises. They were applied in the morning and evening for 2 weeks by the instructions. The BSES and EPDS score of both groups were evaluated in the 1st and 2nd-week follow-up.

DETAILED DESCRIPTION:
With preterm birth, some medical and neurophysiological problems occur in the baby. The mother-father-infant interactions of these babies, who need more intensive care support after birth, are negatively affected by this process. The mother whose baby is in intensive care is separated from her baby and is worried for her life because her baby is underdeveloped and has frequent health problems. All these experiences may cause the mother to lose her maternal role. Therefore, mothers; They may experience a range of negative emotions such as sadness, mourning, fear, grief, disappointment, anger and helplessness, as well as significant psychological disturbances such as postpartum depression and anxiety disorders.

Therefore, appropriate interventions are necessary for early diagnosis and reduction of depression in the postpartum period. Stress-reducing practices such as PMR to be applied to the mother can reduce the mother's anxiety and depression levels, as well as increase breastfeeding self-efficacy. Decrease in depression and increase in breastfeeding self-efficacy will positively affect the mother's breastfeeding and contribute to the growth of the baby.

Participants and sample:

The universe of the study consisted of mothers with preterm infants of 32-36 weeks of gestation who were hospitalized in the NICU.

Sample selection criteria were determined as follows mother's having between 32-36 weeks preterm babies, mother's having enough milk to breastfeed, baby's not having an anomaly that prevents breastfeeding, baby's being fed with breast milk.

To determine the sample size of the study, the power analysis was performed based on a previous study. According to the G*Power analysis result (with a test power of 95% confidence and power of 95.82% for ß: 0.04, alpha: 0.05), the sample size was found to be 70. Considering the possibility of case loss, the total sample size was determined 80 (40 in the experimental group and 40 in the control).

The final number of mothers in the experimental group was 35 and 35 in the control group. As a result, 70 mothers in total were included in the analysis.

Data collecting:

Intervention:

When premature babies were admitted to the NICU, all parents were informed about intensive care settings and premature birth. PMR exercises were applied to the mothers in the experimental group by the researcher and the mothers were given training on the application of the exercises.

Procedure:

Interventions in the experimental group: Introductory information form and EPDS were completed by the mothers before the PMR exercises. PMR exercises were applied to the mothers by the researcher in the milking room (a quiet room) located on the NICU floor and they were given training on the application of the exercises. During the application, it was ensured that only the researcher and the mother were in the room. The application was continued until the mother was able to do the PMR exercises on her own. In case the mother applied the PMR exercises incompletely or incorrectly, the researcher did it to ensure that the mother performed the exercises correctly. It took about 30-45 minutes to do the exercises. After the application and training, the mother was given a guide on the steps of the PMR exercises. The mother was asked to perform the exercises twice a day, in the morning and evening, and record them on the follow-up form. The researcher's contact number was given to the mother for counseling in case she had difficulty following the steps of the PMR exercises. During the follow-ups, the mother was called by the researcher and a message was sent to ensure her continuity in the exercises. At the end of the 1st and 2nd weeks of the follow-up, BSES, EPDS and patient follow-up forms were filled when the mother came for routine controls.

Interventions in the control group: The descriptive information form, BSES and EPDS were first administered to the mothers. BSES and EPDS were applied to the mothers at the end of the 1st and 2nd weeks of follow-up. At the end of the 2nd week, mothers were told how to perform PMR exercises and instructions on PMR exercises were given.

Measurements:

Information Form:

In this form, there are 8 questions about the sociodemographic characteristics of the mother, her working status during pregnancy, the mode of delivery, her participation in the care of the baby in the hospital, the breastfeeding status of the previous baby and the support status of the mother, and the care of the baby after discharge.

Edinburgh Postpartum Depression Scale (EDPS):

It was defined by Cox et al. in 1987 and has been accepted all over the world as a tool that can be used in the recognition of postpartum depression by proving its validity and reliability in many countries, in different languages, until today. It is reported that it can be used for (one) routine screening in all women who have given birth. Validity studies were conducted in 2 separate studies in Turkey, and it is reported that when the cut-off score is 12-13, it is more sensitive in detecting people with true depressive symptoms. The Edinburgh Postpartum Depression Scale is not a diagnostic scale, it is used for symptom screening. The diagnosis needs to be confirmed by clinical examination. The Edinburgh Postpartum Depression Scale is a scale consisting of 10 questions, each of which asks the mother to report how she has felt over the past week by ticking one of four different options. The total score is calculated by giving a score between 0-3 for each item. In some items, the harshest responses are placed at the beginning, while in others they are placed at the end. The score varies between 0-30.

Postpartum Breastfeeding Self-Efficacy Scale (BSES):

It is a 33-item scale developed by Dennis and Faux in 1999 to evaluate mothers' breastfeeding self-efficacy levels. Later, in 2003, a 14-item short form of the scale was developed. The Breastfeeding Self-Efficacy Short Form is a 5-point Likert-type scale (1 = "I'm not sure at all" and 5 = "I'm always sure"). The lowest score that can be obtained from the scale is 14, and the highest score is 70. The higher the score, the higher the breastfeeding self-efficacy. The Turkish validity and reliability study of the scale was carried out by Alus Tokat and Okumuş in 2009.

Patient Follow-up Form:

It was created to track whether mothers of premature infants performing PMR did this exercise twice a day, morning and evening, for a month.

Practice and Guidelines for Progressive Muscle Relaxation (PMR) Exercises:

Before collecting data, one of the researchers received training and certification from a psychotherapist who is an expert in this field in order to be able to perform the PMR exercises. Guidelines for PMR exercises have been prepared in line with the literature and the training received by the researcher. In the guidelines, the person is asked to be in a comfortable place and position, to reach the face by following the large muscle groups gradually, starting from the feet, to tense the muscles in each step, and then to release them. It is necessary to take a deep breath after each muscle group, to stop for a while, and release it slowly.

ELIGIBILITY:
Inclusion Criteria:

* Mother's delivery of a premature baby between 32 weeks-36 weeks + 6 days,
* The mother has enough milk to breastfeed
* The mother's baby does not have an anomaly that prevents breastfeeding,
* Feeding the mother's baby with breast milk

Exclusion Criteria:

* Mothers with babies born outside the range of 32 weeks-36 weeks + 6 days
* Having a baby with a congenital anomaly
* Feeding a mother's baby with a formula other than breast milk

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Enrollment: 70 (Actual)
Dates: Start 2018-11-20 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Breastfeeding Self-Efficacy Scale Score (BSES) | In the 2nd week of follow-up
  BSES score is in the range of 14-70 points, and as the total score increases, breastfeeding self-efficacy also increases.

SECONDARY OUTCOMES:
Edinburgh Postpartum Depression Scale Score (EDPS) | At the end of the 1st and 2nd week of the intervention
  The total score to be taken from this scale varies between 0-30 points. As the total score obtained from the scale increases, the postpartum depression symptoms of the individual increase.
Edinburgh Postpartum Depression Scale (EDPS) Scores Change in Experimental and Control Group | At the end of the 2nd week of follow-up
Edinburgh Postpartum Depression Scale Scores Differences (EDPS) of the Groups | At the end of the 2nd week of follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Birsen Mutlu, Ph.d, Principal Investigator — Istanbul University - Cerrahpasa
Locations (1):
- Kadriye Şahin, Istanbul, Şişli, Turkey (Türkiye)

REFERENCES:
- [Background] Ionio C, Colombo C, Brazzoduro V, Mascheroni E, Confalonieri E, Castoldi F, Lista G. Mothers and Fathers in NICU: The Impact of Preterm Birth on Parental Distress. Eur J Psychol. 2016 Nov 18;12(4):604-621. doi: 10.5964/ejop.v12i4.1093. eCollection 2016 Nov. PMID 27872669
- [Background] Miles MS, Funk SG, Kasper MA. The stress response of mothers and fathers of preterm infants. Res Nurs Health. 1992 Aug;15(4):261-9. doi: 10.1002/nur.4770150405. PMID 1496151
- [Background] Howe TH, Sheu CF, Wang TN, Hsu YW. Parenting stress in families with very low birth weight preterm infants in early infancy. Res Dev Disabil. 2014 Jul;35(7):1748-56. doi: 10.1016/j.ridd.2014.02.015. Epub 2014 Mar 19. PMID 24656293
- [Background] Holditch-Davis D, Santos H, Levy J, White-Traut R, O'Shea TM, Geraldo V, David R. Patterns of psychological distress in mothers of preterm infants. Infant Behav Dev. 2015 Nov;41:154-63. doi: 10.1016/j.infbeh.2015.10.004. Epub 2015 Oct 22. PMID 26495909
- [Background] Henderson J, Carson C, Redshaw M. Impact of preterm birth on maternal well-being and women's perceptions of their baby: a population-based survey. BMJ Open. 2016 Oct 8;6(10):e012676. doi: 10.1136/bmjopen-2016-012676. PMID 27855105
- [Background] Vigod SN, Villegas L, Dennis CL, Ross LE. Prevalence and risk factors for postpartum depression among women with preterm and low-birth-weight infants: a systematic review. BJOG. 2010 Apr;117(5):540-50. doi: 10.1111/j.1471-0528.2009.02493.x. Epub 2010 Jan 29. PMID 20121831
- [Background] Ranger A, Helmert E, Bott TS, Ostermann T, Als H, Bassler D, Hautzinger M, Vagedes J. Physiological and emotional effects of pentatonic live music played for preterm neonates and their mothers in the Newborn Intensive Care Unit: A randomized controlled trial. Complement Ther Med. 2018 Dec;41:240-246. doi: 10.1016/j.ctim.2018.07.009. Epub 2018 Aug 1. PMID 30477847
- [Background] Glover V. Prenatal stress and its effects on the fetus and the child: possible underlying biological mechanisms. Adv Neurobiol. 2015;10:269-83. doi: 10.1007/978-1-4939-1372-5_13. PMID 25287545
- [Background] Simpson M, Schmied V, Dickson C, Dahlen HG. Postnatal post-traumatic stress: An integrative review. Women Birth. 2018 Oct;31(5):367-379. doi: 10.1016/j.wombi.2017.12.003. Epub 2018 Jan 11. PMID 29337007
- [Background] Sharmin KN, Sarwar N, Mumu SJ, Taleb DA, Flora MS. Postnatal depression and infant growth in an urban area of Bangladesh. Midwifery. 2019 Jul;74:57-67. doi: 10.1016/j.midw.2019.03.014. Epub 2019 Mar 22. PMID 30927633
- [Background] Dennis CL. Identifying predictors of breastfeeding self-efficacy in the immediate postpartum period. Res Nurs Health. 2006 Aug;29(4):256-68. doi: 10.1002/nur.20140. PMID 16847899
- [Background] Chuang LL, Lin LC, Cheng PJ, Chen CH, Wu SC, Chang CL. Effects of a relaxation training programme on immediate and prolonged stress responses in women with preterm labour. J Adv Nurs. 2012 Jan;68(1):170-80. doi: 10.1111/j.1365-2648.2011.05765.x. Epub 2011 Jul 20. PMID 21771042
- [Background] Zubaran C, Foresti K. The correlation between breastfeeding self-efficacy and maternal postpartum depression in southern Brazil. Sex Reprod Healthc. 2013 Mar;4(1):9-15. doi: 10.1016/j.srhc.2012.12.001. Epub 2012 Dec 20. PMID 23427927
- [Background] Özcan N, Karagözoğlu Ş. Effects of progressive muscle relaxation exercise, cold application and local anesthesia performed before chest tube removal on pain and comfort levels and vital sings of the patient. Turkiye Klin J Med Sci. 2020;40(3):285-96.
- [Background] Engindeniz A, Küey L, Kültür S. Turkish form of Edinburgh postpartum depression scale validity and reliability study. In: Bahar Sempozyumları 1 Kitabı [Internet]. Ankara: Publications of the Psychiatric Association; 1996 [cited 2022 Feb 11]. p. 51-2. Available from: https://toad.halileksi.net/olcek/edinburgh-dogum-sonrasi-depresyon-olcegi
- [Background] Lawrence RM, Lawrence RA. Breastfeeding: more than just good nutrition. Pediatr Rev. 2011 Jul;32(7):267-80. doi: 10.1542/pir.32-7-267. No abstract available. PMID 21724901
- [Background] Alus Tokat M, Okumus H, Dennis CL. Translation and psychometric assessment of the Breast-feeding Self-Efficacy Scale-Short Form among pregnant and postnatal women in Turkey. Midwifery. 2010 Feb;26(1):101-8. doi: 10.1016/j.midw.2008.04.002. Epub 2008 Jun 9. PMID 18541350
- [Background] Cox JL, Holden JM, Sagovsky R. Detection of postnatal depression. Development of the 10-item Edinburgh Postnatal Depression Scale. Br J Psychiatry. 1987 Jun;150:782-6. doi: 10.1192/bjp.150.6.782. PMID 3651732
- [Background] Helmer G. Progressive Muskelrelaxation nach Edmund Jacobson. In: Burnout und Stress. Springer; 2008. p. 91-110.
- [Background] McCallie MS, Blum CM, Hood CJ. Progressive muscle relaxation. J Hum Behav Soc Environ [Internet]. 2006 Jul 13 [cited 2022 Feb 11];13(3):51-66. Available from: /record/2007-02269-004